CLINICAL TRIAL: NCT03138304
Title: Trial of a Video Game Intervention to Recalibrate Physician Heuristics: A Followup Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Deepika Mohan, Assistant professor of critical care medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOD16070572-03 / PRO16070572
Record Dates: First submitted 2017-04-30; First posted 2017-05-03 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Wounds and Injuries
Keywords: decision making; heuristics
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Group assignment will be masked at the analysis phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adventure video game (Experimental): Night Shift is an adventure video game with the transformational goal of teaching physicians key characteristics of patients with non-representative severe injuries - injuries classified by the American College of Surgeons as life-threatening or critical but that do not fit the archetype of injuries typically requiring treatment at a trauma center. Players take on the persona of Andy Jordan, a young emergency physician who moves home after the disappearance of his estranged grandfather (Robert Jordan) and takes up a job in the local Emergency Department (ED). In the preamble, players learn they have two explicit objectives. First, they must diagnose and treat patients who present to their ED. Second they must solve the mystery of Robert's disappearance: was he murdered or has he simply chosen to disappear?
  Interventions: Behavioral: Video game
- Educational Program (Active Comparator): The educational module consists of two separate apps, both commercially available. myATLS includes a review of each chapter of the Advanced Trauma Life Support (ATLS) textbook, a series of videos demonstrating common trauma procedures, and clinical resources including checklists for use at the bedside. Trauma Life Support MCQ Review includes 550 multiple-choice questions with correct answers and explanations. The investigators will ask physicians to review the myATLS app and then complete questions in the Trauma Life Support MCQ Review, spending at least 1 hour on the combined tasks.
  Interventions: Behavioral: Educational program

INTERVENTIONS:
Behavioral: Video game — Night Shift is an adventure video game with the transformational goal of teaching physicians key characteristics of patients with non-representative severe injuries - injuries classified by the American College of Surgeons as life-threatening or critical but that do not fit the archetype of injuries typically requiring treatment at a trauma center.
  Arms: Adventure video game
Behavioral: Educational program — Two commercially available applications designed to teach physicians the trauma triage guidelines disseminated by the American College of Surgeons.
  Arms: Educational Program

SUMMARY:
The objective of this study is to measure the duration of two different types of interventions to change physician decision making in trauma triage: a video game and an educational program.

DETAILED DESCRIPTION:
Treatment at trauma centers improves outcomes for patients with moderate-to-severe injuries. Accordingly, professional organizations, state authorities, and the federal government have endorsed the systematic triage and transfer of these patients to trauma centers either directly from the field or after evaluation at a non-trauma center. Nonetheless, between 30 to 40% of patients with moderate-to-severe injuries still only receive treatment at non-trauma centers, so-called under-triage. Most of this under-triage occurs because of physician decisions (rather than first-responder decisions). Existing efforts to change physician decision making focus primarily on knowledge of clinical practice guidelines and attitudes towards the guidelines. These strategies ignores the growing consensus that decision making reflects both knowledge as well as intuitive judgments (heuristics). Heuristics, mental short cuts based on pattern recognition, drive the majority of decision making. The investigators developed an adventure video game (Night Shift) to serve as a novel method of recalibrating physician heuristics in trauma triage and compared its efficacy with a standard educational program. This study is designed to measure the degradation of the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Physicians who care for adult patients in the Emergency Department.
* Physicians who work at a non-trauma center.
* Physicians who work at a Level III/IV trauma center.

Exclusion Criteria:

* Physicians who work only at a Level I/II trauma center.
* Physicians who do not practice in the US.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Undertriage | 6 months after completion of the intervention
  Physicians in both arms of the study will be asked to complete an outcome assessment tool - a virtual simulation - six months after completion of their intervention. The virtual simulation replicates the environment of the ED. Physicians have to manage 10 patients that appear concurrently, while also responding to a series of audio-visual distractors. Specifically, they must provide information on whether they will admit, transfer, or discharge the patients home. The investigators will calculate an under-triage rate for each physician (the number of simulated patients with severe injuries not transferred to a trauma center), will summarize the under-triage rate by group (Night Shift v. educational control), and will assess the difference in those rates.

SECONDARY OUTCOMES:
Undertriage for nonrepresentative and representative injuries | 6 months after completion of the intervention
  We will categorize severely injured patients on the virtual simulation (the outcome assessment tool) as having representative or non-representative injuries. We will summarize the undertriage rate of representative/non-representative injuries by intervention, and will compare the difference in those rates between groups.
Degradation in treatment effect | 6 months after completion of the intervention.
  We will compare the undertriage rate of physicians the first and second time they complete the virtual simulation (time zero = initial enrollment; time one = six months post intervention). We will compare the difference in the undertriage rates by intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Mohan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers may contact the PI for access to deidentified participant data. It will be released conditional on IRB approval.

REFERENCES:
- [Derived] Mohan D, Farris C, Fischhoff B, Rosengart MR, Angus DC, Yealy DM, Wallace DJ, Barnato AE. Efficacy of educational video game versus traditional educational apps at improving physician decision making in trauma triage: randomized controlled trial. BMJ. 2017 Dec 12;359:j5416. doi: 10.1136/bmj.j5416. PMID 29233854